CLINICAL TRIAL: NCT02578199
Title: Novel and Scalable Internet Supplemented Weight Loss Treatment in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1106008713-B; R03DK104008-01 (NIH)
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2016-11

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Motivational Interviewing; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- motivational interviewing and nutrition (Experimental): Motivational interviewing and nutritional counseling.
  Interventions: Behavioral: motivational interviewing and nutrition

INTERVENTIONS:
Behavioral: motivational interviewing and nutrition — Motivational Interviewing and Nutritional Counseling

SUMMARY:
Motivational interviewing and nutritional counseling for weight loss in primary care.

DETAILED DESCRIPTION:
Overweight and obese participants will be recruited through local primary care offices. This study will test the effectiveness of motivational interviewing and nutritional counseling for weight loss. The treatment will be supplemented by internet support.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-55
* Daily access to internet and phone
* Recruited through local primary care offices.
* Age 18-65

Exclusion Criteria:

* Co-existing physical and/or psychiatric conditions that require more significant treatment (e.g., bipolar disorder, psychotic illnesses), and/or require more intensive treatment or hospitalization (e.g., suicidality, severe mood disorders)
* Meets criteria for current substance abuse/dependence
* Currently receiving psychiatric, psychological, behavioral, or pharmacologic treatment that is known to affect weight or eating
* Pregnant, breastfeeding, or plans to become pregnant during the treatment period
* Cardiac disease, including ischemic heart disease, congestive heart failure, conduction abnormalities, or a history of heart attack
* Serious neurologic illnesses (e.g., seizure history) or medical illnesses (e.g., impaired hepatic or renal function)
* Uncontrolled diabetes, thyroid conditions, or hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-02 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Barnes, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Barnes RD, Ivezaj V, Martino S, Pittman BP, Paris M, Grilo CM. 12 Months later: Motivational interviewing plus nutrition psychoeducation for weight loss in primary care. Eat Weight Disord. 2021 Aug;26(6):2077-2081. doi: 10.1007/s40519-020-00994-5. Epub 2020 Sep 7. PMID 32894453
- [Derived] Barnes RD, Ivezaj V, Martino S, Pittman BP, Paris M, Grilo CM. Examining motivational interviewing plus nutrition psychoeducation for weight loss in primary care. J Psychosom Res. 2018 Jan;104:101-107. doi: 10.1016/j.jpsychores.2017.11.013. Epub 2017 Nov 28. PMID 29275778
- [Derived] Barnes RD, Ivezaj V, Martino S, Pittman BP, Grilo CM. Back to Basics? No Weight Loss from Motivational Interviewing Compared to Nutrition Psychoeducation at One-Year Follow-Up. Obesity (Silver Spring). 2017 Dec;25(12):2074-2078. doi: 10.1002/oby.21972. Epub 2017 Oct 31. PMID 29086484

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing and Nutrition
Started | 31
Completed | 27
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Motivational Interviewing and Nutrition
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 16
  More than one race | 1
  Unknown or Not Reported | 2
Baseline Weight [Mean (Standard Deviation); unit: pounds] | 212.2 (34.0)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight in Pounds
Description: Body weight in pounds measured 3 months after starting treatment.
Time Frame: 3 months
Population: 27 participants completed treatment, 28 participants completed the post treatment assessment (i.e., one participant who dropped from treatment completed the post treatment assessment).
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Motivational Interviewing and Nutrition
Number analyzed (Participants) | 28
pounds | 207.4 (32.7)

2. Secondary Outcome: Body Weight in Pounds
Description: Body weight in pounds measured 6 months after starting treatment (3 month follow-up after active treatment ends).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Motivational Interviewing and Nutrition
Number analyzed (Participants) | 27
pounds | 204.8 (34.6)

ADVERSE EVENTS:
Arm/Group | Motivational Interviewing and Nutrition
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes